CLINICAL TRIAL: NCT06591403
Title: INVESTIGATION OF PERIPHERAL OXYGEN SATURATION VALUES MEASURED IN DIFFERENT BODY POSITIONS AND FINGERS
Brief Title: INVESTIGATION OF PERIPHERAL OXYGEN SATURATION VALUES MEASURED IN DIFFERENT BODY POSITIONS AND FINGERS IN HEALTHY YOUNG ADULT INDIVIDUALS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uludag University (Other)
Responsible Party: Principal Investigator, Dilek Yilmaz, PhD, Associate Professor, Uludag University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2023-25/25
Record Dates: First submitted 2024-09-07; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Peripheral Oxygen Saturation; Healthy Individuals
Keywords: Body Positions; Oxygenation; Pulse Oximetry

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- the different body positions and fingers (Experimental)
  Interventions: Other: the index and middle fingers of each participant's active hand

INTERVENTIONS:
Other: the index and middle fingers of each participant's active hand — A pulse oximeter was placed simultaneously on the index and middle fingers of each participants active hand while they were in an upright sitting position. After the pulse oximeter was placed on both fingers for one minute, stable values seen on its screen for at least three seconds were recorded. Then, the participants were placed in a supine position, and after a 10-minute rest, similar measurements were repeated with a pulse oximeter placed on the index and middle fingers of the active hand.

SUMMARY:
This study aims to examine peripheral oxygen saturation values measured in different body positions and fingers in healthy young adult individuals.

The research was planned in a quasi-experimental design. The research population consisted of students/healthy young adults studying at Bursa Uludağ University Faculty of Health Sciences between January 2024 and May 2024. The research sample consisted of a total of 200 volunteer individuals who met the research limitations.

The research data were collected using the Individual Introduction Form and Peripheral Oxygen Saturation Monitoring Form. A pulse oximeter was placed simultaneously on the index and middle fingers of each participant's active hand while they were in an upright sitting position. After the pulse oximeter was placed on both fingers for one minute, stable values seen on its screen for at least three seconds were recorded. Then, the participants were placed in a supine position, and after a 10-minute rest, similar measurements were repeated with a pulse oximeter placed on the index and middle fingers of the active hand.

ELIGIBILITY:
Inclusion Criteria:

* participating voluntarily in the study
* being aged over 18 years
* not having any acute or chronic disease

Exclusion Criteria:

* being less than 18 years of age,
* having anemia,
* not wanting to participate in the study, or during the course of the research, wishing to withdraw from the study,
* having an oxygen saturation value of less than 90%,
* being unable to tolerate a 0° prone position (bradycardic).

Ages: 19 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 200 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-01-20 (Actual); Study Completion 2024-05-15 (Actual)

PRIMARY OUTCOMES:
heart rate | 5 months
  heart rate in beats
peripheral oxygen saturation | 5 months
  peripheral oxygen saturation in percentage

SECONDARY OUTCOMES:
weight | 5 months
  weight in kilograms
height | 5 months
  height in meters

CONTACTS AND LOCATIONS:
Locations (1):
- Bursa Uludag University Faculty of Health Sciences, Bursa, Nilüfer, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided